CLINICAL TRIAL: NCT01324141
Title: A Pilot Trial Assessing the Feasibility of Delivering Topical MTS-01 to Reduce Dermatitis in Patients Receiving Intensity Modulated Radiation With Concurrent 5-Fluorouracil and Mitomycin-C for Stage I-III Carcinoma of the Anal Canal
Brief Title: Topical MTS-01 for Dermatitis During Radiation and Chemotherapy for Anal Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow, insufficient accrual and failure to meet endpoints.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Deborah Citrin, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110129; 11-C-0129
Record Dates: First submitted 2011-03-25; First posted 2011-03-28 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-10

CONDITIONS: Anal Cancer
Keywords: Anal Cancer; Radioprotector; Topical; Radiation; Dermatitis
MeSH Terms: conditions — Anus Neoplasms; Dermatitis | interventions — tempol; Fluorouracil; Mitomycin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1/Chemo + Radiation (Experimental): Chemo + Radiation
  Interventions: Drug: Tempol; Drug: 5-Fluorouracil; Drug: Mitomycin-C; Procedure: Radiation Therapy

INTERVENTIONS:
Drug: Tempol — Tempol gel will be applied to the bilateral groins and the gluteal cleft, avoiding a 3 cm radius from the anal verge, immediately prior to each fraction of radiation therapy (RT).
  Other Names: MBM-02
Drug: 5-Fluorouracil — 5-FU will be delivered as 1000mg/m(2)/day as 96 hour continuous infusion beginning on day 1 and 29.
  Other Names: 5-FU
Drug: Mitomycin-C — Mitomycin-C (MMC) will be delivered at a dose of 10mg/m(2) on days 1 and 29
  Other Names: MMC
Procedure: Radiation Therapy — Radiation therapy (RT) will be delivered to a total dose of 50-54 Gray (Gy) based on tumor characteristics.
  Other Names: RT

SUMMARY:
Background:

- Radiation and chemotherapy treatments for anal cancer can cause irritation of the skin that can lead to redness and tenderness, and in some cases can be so severe that it results in blistering or peeling of the skin during treatment. These conditions cause discomfort and may require breaks from radiation treatment. Researchers are interested in determining whether MTS-01, a drug that protects cells and tissues from the effects of radiation, can be given before radiation treatment to prevent these side effects and reduce the irritation of the skin during chemotherapy and radiation for anal cancer.

Objectives:

- To determine the safety and effectiveness of topical MTS-01 given before radiation in the groin and gluteal cleft of patients receiving combined radiation and chemotherapy for anal cancer.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with cancer of the anal canal and are eligible to receive radiation and chemotherapy treatments.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, imaging studies and physical examination of the anal canal, and biopsies as needed to evaluate eligibility for treatment.
* Participants will be scheduled for radiation and chemotherapy treatments on the following schedule:
* Radiation given 5 days per week for 6 weeks, with topical MTS-01 treatment on the skin in the groin areas and between the buttocks before each treatment
* Mitomycin C given intravenously on days 1 and 29 of treatment
* 5-Fluorouracil given intravenously over 4 days (first week and fifth week) during radiation treatment
* Participants will be monitored throughout the treatment for side effects, with photographs of the treatment area and frequent blood tests.
* Following the end of radiation, participants will have followup visits for 1 year with blood tests and imaging studies to evaluate the response to treatment.

DETAILED DESCRIPTION:
Background:

* Patients with non-metastatic carcinoma of the anal canal are treated with concurrent mitomycin C (MMC), 5-fluorouracil (5-FU), and radiotherapy (RT) in the curative setting in an attempt to preserve the anal sphincter.
* Radiation dermatitis is a uniform complication of this therapy which frequently results in treatment delay due to pain and discomfort. High grade dermatitis may also become superinfected in the setting of decreased blood counts from chemotherapy and diarrhea from radiation proctitis, further delaying therapy. Approaches that decrease toxicity may be particularly important in patients infected with human immunodeficiency virus (HIV).
* MTS-01 (tempol, 4-hydroxy-2,2,6,6-tetramethylpiperidine-1-oxyl) is a piperidine nitroxide known to act as a chemical radioprotector with selective protection of normal versus tumor tissue.
* Tempol gel (tempol 70 mg/mL plus water, ethanol, and hydroxypropyl cellulose) has been evaluated as a topical radioprotector in pilot trials that included a variety of sites.

Objectives:

* Primary Objective: To determine the safety and tolerability of topical MTS-01 on a daily basis prior to irradiation in the groin and gluteal cleft of patients receiving combined therapy with MMC, 5-FU, and RT for carcinoma of the anal canal.
* Secondary Objectives will include evaluation of the following endpoints in a preliminary fashion:

  * To describe the rates and severity of skin toxicity in patients treated with this regimen
  * To describe the need for toxicity related treatment breaks with this regimen
  * To describe the opiate requirements in patients treated with this regimen
  * To describe 12-month progression-free survival, disease-free survival, and overall survival in patients treated with concurrent chemotherapy, radiation therapy, and MTS-01
  * Evaluate the effects of antiretroviral therapy, 5-fluorouracil, mitomycin C, and radiation on low level persistent HIV viremia and HIV genetic diversity during therapy and recovery
  * To evaluate the feasibility of collecting HIV ribonucleic acid (RNA) and mononuclear cells from rectal associated lymphoid tissue for correlative studies
  * Collect and store anal cytology and core needle biopsies of tumor for future human papillomavirus infection (HPV) and tumor based analyses

Eligibility:

* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2.
* Histologically confirmed carcinoma of the anal canal without evidence of distant metastases
* No contraindications to definitive chemoradiotherapy for carcinoma of the anal canal

Design:

This is a pilot trial of topical MTS-01 in patients receiving MMC, 5-FU, and intensity-modulated radiation therapy (IMRT) for definitive management of carcinoma of the anal canal. Fifteen patients will be enrolled. MMC will be delivered at a dose of 10mg/m(2) on days 1 and 29. 5-FU will be delivered as 1000mg/m(2)/day as 96 hour continuous infusion beginning on day 1 and 29. RT will be delivered to a total dose of 50-54 Gy based on tumor characteristics. Tempol gel will be applied to the bilateral groins and the gluteal cleft, avoiding a 3 cm radius from the anal verge, immediately prior to each fraction of RT. Radiation Therapy Oncology Group (RTOG) grading will be used to evaluate skin toxicity in both the groin and gluteal cleft weekly during treatment and at 4 weeks, 3 months and 6 months after completion of treatment. The duration of treatment, number of treatment breaks, opiate requirements, and level of pain will be evaluated weekly during treatment and at 4 weeks and 3 months after the completion of treatment. Disease control will be assessed at 4 weeks, 3 months, 6 months, 9 months, and 12 months of follow-up.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically proven, invasive primary squamous, basaloid, or cloacogenic carcinoma of the anal canal, stage T1-4, N0-3
* No previous therapy for anal cancer.
* Age greater than or equal to 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate bone marrow, renal, and hepatic function defined as

  * Absolute neutrophil count greater than or equal to 1,000 cells/mm(3)
  * Platelet count greater than or equal to 100,000/mm(3)
  * Hemoglobin greater than or equal to 8mg/dL
  * Creatinine clearance > 60 mL/min using Cockcroft-Gault formula
  * Bilirubin less than or equal to 1.5 times upper limit of normal (ULN) unless, during screening, the patient is receiving protease inhibitor therapy (i.e. indinavir, ritonavir, nelfinavir, and atazanavir) known to be associated with increased bilirubin: in this case total bilirubin less than or equal to 7.5 mg/dl and the direct fraction is less than or equal to 0.7 mg/dl.
  * White blood cell (WBC) greater than or equal to 3,000/microL
  * Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than or equal to 3 times the upper limit of normal
  * International normalized ratio (INR) less than or equal to 1.5
* Patients of childbearing potential must be willing to use a medically effective means of birth control for the duration of treatment and six weeks after treatment.
* Patients must be willing and able to provide informed consent

EXCLUSION CRITERIA:

* Contraindications to radiotherapy such as a history of prior radiotherapy to the pelvis or a history of inflammatory bowel disease
* Prior malignancy except:

  * non-melanoma skin cancer
  * controlled Kaposi's Sarcoma (no chemotherapy for KS for 3 months, and no expected need for chemotherapy for the 12-month period of the study)
  * other malignancies with disease free period of at least 3 years
* Presence of metastatic disease (M1)
* Co-morbidity that in the estimation of the principal investigator would make the patient unable to tolerate treatment
* Pregnant or lactating females
* Human immunodeficiency virus (HIV) positive patients with cluster of differentiation 4 (CD4) < 100 cells/mL AND ECOG performance status (PS) greater than 2.
* Dermatitis in the anticipated radiation treatment portal.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2011-03-18 (Actual); Primary Completion 2015-04-15 (Actual); Study Completion 2015-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah E Citrin, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Thun MJ. Cancer statistics, 2009. CA Cancer J Clin. 2009 Jul-Aug;59(4):225-49. doi: 10.3322/caac.20006. Epub 2009 May 27. PMID 19474385
- [Background] Bower M, Powles T, Newsom-Davis T, Thirlwell C, Stebbing J, Mandalia S, Nelson M, Gazzard B. HIV-associated anal cancer: has highly active antiretroviral therapy reduced the incidence or improved the outcome? J Acquir Immune Defic Syndr. 2004 Dec 15;37(5):1563-5. doi: 10.1097/00126334-200412150-00004. PMID 15577408
- [Background] Crum-Cianflone NF, Hullsiek KH, Marconi VC, Ganesan A, Weintrob A, Barthel RV, Agan BK; Infectious Disease Clinical Research Program HIV Working Group. Anal cancers among HIV-infected persons: HAART is not slowing rising incidence. AIDS. 2010 Feb 20;24(4):535-43. doi: 10.1097/QAD.0b013e328331f6e2. PMID 19926961

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1/Chemo + Radiation
Started | 6
Completed | 4
Not Completed | 2
Not completed — Declined to participate before treatment started | 1
Not completed — Disease progression on study | 1

BASELINE CHARACTERISTICS:
Population: Some baseline data was captured for 1/6 participants that later withdrew before treatment.
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.85 (5.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG 0 is asymptomatic. ECOG 1 is symptomatic but ambulatory. ECOG 2 is <50% in bed. ECOG 3 is >50% in bed. ECOG 4 is bedbound. ECOG 5 is death. ECOG was not captured for one participant that withdrew before treatment. Population: ECOG data was not captured for 1/6 participants that withdrew before treatment.
  Participants
    ECOG 0: number analyzed (Participants) | 5
    ECOG 0 | 3
    ECOG 1: number analyzed (Participants) | 5
    ECOG 1 | 2
    ECOG 2: number analyzed (Participants) | 5
    ECOG 2 | 0
    ECOG3: number analyzed (Participants) | 5
    ECOG3 | 0
    ECOG4: number analyzed (Participants) | 5
    ECOG4 | 0
    ECOG 5: number analyzed (Participants) | 5
    ECOG 5 | 0
Human Immunodeficiency Virus (HIV) Status [Count of Participants; unit: Participants] — HIV is a virus that attacks the body's immune system that can lead to serious illness and/or death.
  HIV positive = HIV test detected HIV in blood or saliva sample HIV negative = HIV test did not detect HIV in blood or saliva sample Population: HIV status was not captured for 1/6 participants that withdrew before treatment.
  Participants
    HIV Positive: number analyzed (Participants) | 5
    HIV Positive | 1
    HIV Negative: number analyzed (Participants) | 5
    HIV Negative | 4
Human Papilloma Status (Anal Swab) [Count of Participants; unit: Participants] — HPV is a sexually transmitted infection that can cause warts and cervical cancer.
  HPV positive = HPV test detects deoxyribonucleic acid (DNA) or ribonucleic acid (RNA) of HPV in cell sample HPV negative = HPV did not detect DNA or RNA of HPV in cell sample Population: HPV status was not captured for 1/6 participants that withdrew before treatment.
  Participants
    HPV Positive: number analyzed (Participants) | 5
    HPV Positive | 0
    HPV Negative: number analyzed (Participants) | 5
    HPV Negative | 5
T Stage [Count of Participants; unit: Participants] — T Stage was measured by the American Joint Committee on Cancer (AJCC 7th Edition).
  T = tumor/describes size of original tumor T1-4 is increasing size and/or local extension of the primary tumor. Population: T Stage was not captured for 1/6 participants that withdrew before treatment.
  Participants
    T1: number analyzed (Participants) | 5
    T1 | 0
    T2: number analyzed (Participants) | 5
    T2 | 2
    T3: number analyzed (Participants) | 5
    T3 | 3
    T4: number analyzed (Participants) | 5
    T4 | 0
N Stage [Count of Participants; unit: Participants] — N Stage was measured by the Stage American Joint Committee on Cancer (AJCC 7th Edition) N = node/cancer present in lymph nodes N0 = no lymph node metastases N1 = cancer spread to groin, rectum, and pelvic or external iliac nodes N2 = Metastasis in unilateral internal iliac and/or unilateral inguinal lymph node N3 = Metastasis in perirectal and inguinal lymph nodes and/or bilateral internal iliac and/or bilateral inguinal lymph nodes Population: N Stage was not captured for 1/6 participants that withdrew before treatment.
  Participants
    N0: number analyzed (Participants) | 5
    N0 | 4
    N1: number analyzed (Participants) | 5
    N1 | 0
    N2: number analyzed (Participants) | 5
    N2 | 0
    N3: number analyzed (Participants) | 5
    N3 | 1
Stage [Count of Participants; unit: Participants] — Stage was measured by the American Joint Committee on Cancer (AJCC 7th Edition) Stage I - cancer has spread beyond to layer of anal tissue Stage II - tumor >2cm Stage III - cancer is any size but has not grown into nearby organs, or has spread into nearby organs Stage IV- most advanced stage of cancer; cancer is any size and may/may not have spread to nearby organs Stage V - Population: Stage was not captured for 1/6 participants that withdrew before treatment.
  Participants
    I: number analyzed (Participants) | 5
    I | 0
    II: number analyzed (Participants) | 5
    II | 4
    IIIA: number analyzed (Participants) | 5
    IIIA | 0
    IIIB: number analyzed (Participants) | 5
    IIIB | 1
    IV: number analyzed (Participants) | 5
    IV | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 1 and Higher Adverse Events Possibly, Probably, or Definitely Related to Topical MTS-01 and 5-Fluoruracil (5-FU)/Mitomycin C (MMC)/Intensity-modulated Radiotherapy (IMRT)
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v4.0. Grade 1 is mild, Grade 2 is moderate, Grade 3 is severe, Grade 4 is life threatening, and Grade 5 is death related to adverse event.
Time Frame: Date treatment consent signed to date off study, approximately, 36 months and 10 days.
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Number; unit: Adverse events
Groups:
- MTS-01 Grade 1: Grade 1 is mild adverse events.
- MTS-01 Grade 2; 5FU/MMC/IMRT Grade 2: Grade 2 is moderate adverse events.
- MTS-01 Grade 3: Grade 3 is severe adverse events.
- 5-FU/MMC/IMRT Grade 3-4: Grade 3 is severe adverse events and Grade 4 is life threatening adverse events.
Arm/Group | MTS-01 Grade 1 | MTS-01 Grade 2 | MTS-01 Grade 3 | 5FU/MMC/IMRT Grade 2 | 5-FU/MMC/IMRT Grade 3-4
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Adverse events
  Radiation dermatitis | 0 | 0 | 0 | 2 | 3
  Nausea | 0 | 0 | 0 | 3 | 0
  Abdominal pain | 0 | 0 | 0 | 1 | 0
  Diarrhea | 1 | 1 | 0 | 1 | 2
  Gastroesophageal reflux | 0 | 0 | 0 | 1 | 0
  Mucositis | 0 | 0 | 0 | 1 | 0
  Urinary tract pain | 0 | 0 | 0 | 2 | 0
  Bladder spasm | 0 | 0 | 0 | 1 | 0
  Urinary incontinence | 0 | 0 | 0 | 1 | 0
  Fatigue | 1 | 0 | 1 | 1 | 0
  Hypoglycemia | 1 | 0 | 0 | 0 | 0
  Transaminitis | 0 | 0 | 0 | 1 | 0
  Hypoalbuminemia | 0 | 0 | 0 | 1 | 0
  Hypocalcemia | 0 | 0 | 0 | 1 | 0
  Myalgia | 0 | 0 | 0 | 1 | 0
  Headache | 0 | 0 | 0 | 0 | 1
  Syncope | 0 | 0 | 0 | 0 | 1
  Infection | 0 | 0 | 0 | 1 | 1
  Insomnia | 0 | 0 | 0 | 1 | 0
  Pain | 0 | 0 | 0 | 2 | 2
  Leukopenia | 0 | 0 | 0 | 0 | 5
  Lymphopenia | 0 | 0 | 0 | 0 | 5
  Neutropenia | 0 | 0 | 0 | 2 | 3
  Febrile neutropenia | 0 | 0 | 0 | 0 | 1
  Thrombocytopenia | 0 | 0 | 0 | 2 | 0
  Anemia | 0 | 0 | 0 | 3 | 0
  Cluster of Differentiation (CD4) count decrease | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately, 36 months and 10 days.
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 5

3. Secondary Outcome: Mean Grade of Toxicity at Each Timepoint and Location for All Participants Who Underwent Treatment
Description: RTOG grade 1-5 were used to assess skin toxicity in the groin (right and left inguinal area) and gluteal cleft, as well as two control sites. Grade 0 is no skin toxicity, Grade 1 is follicular, faint or dull erythema, Grade 3 is tender or bright erythema, Grade 3 is confluent, moist desquamation, Grade 4 is ulceration, hemorrhage, or necrosis, and Grade 5 is death due to radiation toxicity.
Time Frame: baseline, weeks 1-6, follow up at 1 week, follow up at 2 weeks, and follow up at 4 weeks
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Standard Deviation); unit: Grade
Groups:
- Gluteal Cleft: MTS-01 and 5-Fluoruracil (5-FU)/Mitomycin C (MMC) applied to gluteal cleft. Intensity-modulated Radiotherapy (IMRT) administered.
- Right Inguinal Area: MTS-01 and 5-Fluoruracil (5-FU)/Mitomycin C (MMC) applied to right inguinal area.
  Intensity-modulated Radiotherapy (IMRT) administered.
- Left Inguinal Area: MTS-01 and 5-Fluoruracil (5-FU)/Mitomycin C (MMC) applied to left inguinal area.
  Intensity-modulated Radiotherapy (IMRT) administered.
- Left Inguinal Control (C1): Control site within the treatment area. Radiation only.
- Umbilical Control (C2): Control site outside of the treatment field. MTS-01 only.
Arm/Group | Gluteal Cleft | Right Inguinal Area | Left Inguinal Area | Left Inguinal Control (C1) | Umbilical Control (C2)
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5
Grade
  Baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 1 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Week 3 | 0.4 (0.5) | 0.2 (0.5) | 0.2 (0.5) | 0.2 (0.5) | 0 (0)
  Week 4 | 0.6 (0.5) | 0.6 (0.5) | 0.6 (0.5) | 0.2 (0.5) | 0 (0)
  Week 5 | 1 (0.7) | 0.8 (0.5) | 0.8 (0.5) | 0.2 (0.5) | 0 (0)
  Week 6 | 1.2 (1.1) | 1.2 (0.5) | 1.2 (0.5) | 0.4 (0.5) | 0 (0)
  Follow up at 1 week | 1.8 (0.8) | 1 (0) | 1 (0) | 0.6 (0.5) | 0 (0)
  Follow up at 2 weeks | 1.2 (0.5) | 1 (0) | 1 (0) | 0.8 (0.5) | 0 (0)
  Follow up at 4 weeks | 0.4 (0.5) | 0.2 (0.5) | 0.2 (0.5) | 0.6 (0) | 0 (0)

4. Secondary Outcome: Number of Participants That Required a Treatment Break Relative to Hematologic Toxicity (Non-dermatologic)
Description: Number of participants that required a treatment break relative to hematologic (e.g. thrombocytopenia, leukopenia) toxicity (non-dermatologic).
Time Frame: From beginning until completion of radiation treatment up to 46 days
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 0

5. Secondary Outcome: Number of Participants Treated With Topical MTS-01 and 5-Fluoruracil (5-FU)/Mitomycin C (MMC)/Intensity-modulated Radiotherapy (IMRT) That Required Opiates
Description: Opiates are strong drugs prescribed by prescription used for maximum pain relief.
Time Frame: Completion of study, approximately 14 months after start of treatment
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 5

6. Secondary Outcome: Number of Participants With 12-month Progression-free Survival Treated With 5-Fluoruracil (5-FU)/Mitomycin C (MMC)/Intensity-modulated Radiotherapy (IMRT)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST0 version 1.1. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions.
Time Frame: 12 months
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 4

7. Secondary Outcome: Change in the Levels of Number of Human Immunodeficiency Virus (HIV) in the Circulation Pre and Post Treatment
Description: Change in the levels of number of Human Immunodeficiency Virus (HIV) in the circulation pre and post treatment
Time Frame: Completion of study, approximately 14 months
Population: The participants were screened for HIV before enrollment. Only 1 participant was HIV positive. However, the participant with HIV came off study before post treatment was collected so change cannot be assessed. As pre-specified in the protocol, participants are taken off study for disease progression.
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 0

8. Secondary Outcome: Ratio of the Number of Cluster of Differentiation 4 (CD4): Cluster of Differentiation 8 (CD8) Cells in the Circulation and Tissue Pre and Post Treatment
Description: Ratio of the number Cluster of Differentiation 4 (CD4): Cluster of Differentiation 8 (CD8) cells in the circulation and tissue pre and post treatment. The number of cells of CD4 are divided by the number of cells of CD8.
Time Frame: Pre-treatment and post treatment tissue (CD4), and pre-treatment and post treatment circulation (CD8)
Population: 3/6 participants were analyzed because 1 participant was enrolled but withdrew before treatment, samples were collected at the time of optional biopsy which was conducted in 3 patients.
Measure: Mean (Full Range); unit: Ratio of CD4:CD8 cells
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 3
Ratio of CD4:CD8 cells
  CD4:CD8 Pre-treatment tissue | 5.2 [3.6 to 7.0]
  CD4:CD8 post treatment tissue | 1.89 [0.5 to 3.2]
  CD4:CD8 pre-treatment circulation | 2.95 [2.4 to 3.3]
  CD4:CD8 post treatment circulation | 1.56 [0.9 to 2.1]

9. Secondary Outcome: Number of Participants With 12 Month Disease Free Survival (DFS) Treated With 5-Fluoruracil (5-FU)/Mitomycin C (MMC)/Intensity-modulated Radiotherapy (IMRT)
Description: DFS is defined as the duration of time from start of treatment to time of progression. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST0 version 1.1. Progression is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. And the appearance of one or more new lesions.
Time Frame: 12 months
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 4

10. Secondary Outcome: Overall Survival
Description: OS is defined as the duration of time from start of treatment to time of death.
Time Frame: start of treatment to time of death, approximately 14 months
Population: This outcome measure could not be completed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
months | NA [NA to NA] — The overall survival was to be reported as a median. One participant withdrew. Of the 5 remaining participants, none died while on study, one of these patients was removed from study for progression and was censored at that time.

11. Secondary Outcome: Peripheral Blood Mononuclear Cells (Vascular Endothelial Growth Factor (VEGF), Tumor Necrosis Factor Alpha (TNF-alpha), Interleukin-7 (IL-7), and Transforming Growth Factor Beta-1 (TGF-beta1) Cell Counts at Baseline and Course 1 Day 28
Description: Peripheral blood mononuclear cells (Vascular Endothelial Growth Factor (VEGF), Tumor Necrosis Factor alpha (TNF-alpha), Interleukin-7 (IL-7), and Transforming Growth Factor beta-1 (TGF-beta1) were sampled from peripheral blood from rectal associated lymphoid tissue to evaluate immune cell subsets at baseline and after treatment with MTS-0 and 15-Fluoruracil (5-FU)/Mitomycin C (MMC)/Intensity-modulated Radiotherapy (IMRT). It is unknown if a lower or higher numbers has prognostic significance.
Time Frame: Baseline and Course 1 Day 28
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
pg/ml
  VEGF at baseline | 151.24 (45.0)
  VEGF at Course 1 Day 28 | 127.26 (63.6)
  TNF-alpha at baseline | 3.36 (1.2)
  TNF-alpha at Course 1 Day 28 | 3.21 (2.5)
  IL-7 at baseline | 11.32 (6.2)
  IL-7 at Course 1 Day 28 | 15.62 (10.3)
  TGF-beta 1 at baseline | 14435 (3711.7)
  TGF-beta 1 at Course 1 Day 28 | 7946 (2729.3)

12. Secondary Outcome: Number of Participants With Tumor Tissue Negative for Human Papilloma Virus (HPV)
Description: HPV is a sexually transmitted infection that can cause warts and cervical cancer. HPV test detects deoxyribonucleic acid (DNA) or ribonucleic acid (RNA) of HPV in a cell sample (i.e. cervical).
Time Frame: Pretreatment
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Participants | 5

13. Secondary Outcome: Brief Pain Inventory Score
Description: The Brief Pain Inventory Scale is a questionnaire that asks the participant to rate their pain on a scale of 0 (no pain) to 10 (worst pain).
Time Frame: Baseline, Week 3, Week 6, 1 month follow up, and 3 months follow up
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Scores on a scale
  Worst pain at baseline | 4.8 [0 to 10]
  Worst pain at treatment week 3 | 3.5 [0 to 8]
  Worst pain at treatment week 6 | 7.2 [4 to 10]
  Worst pain at 1 month follow up | 3.1 [0 to 9]
  Worst pain at 3 months follow up | 2.1 [0 to 5]
  Least pain at baseline | 1.4 [0 to 4]
  Least pain at treatment week 3 | 1.5 [0 to 4]
  least pain at treatment week 6 | 3.6 [1 to 5]
  Least pain at 1 month follow up | 1.2 [0 to 3]
  Least pain at 3 months follow up | 2.8 [0 to 5]
  Average pain at baseline | 1.8 [0 to 4]
  Average pain at treatment week 3 | 1.9 [0 to 3.5]
  Average pain at treatment week 6 | 5.0 [2 to 7]
  Average pain at 1 month follow up | 2.0 [0 to 6]
  Average pain at 3 months follow up | 3.0 [0 to 6]
  Pain at time of survey at baseline | 1.6 [0 to 6]
  Pain at time of survey at treatment week 3 | 1.3 [0 to 5]
  Pain at time of survey at treatment week 6 | 5.4 [2 to 9]
  Pain at time of survey a 1 month follow up | 2.2 [0 to 6]
  Pain at time of survey at 3 months follow up | 2.2 [0 to 5]

14. Secondary Outcome: Pain Interference
Description: The Brief Pain Inventory Scale questionnaire were used to assess pain interference. Participants rated pain interference on a scale of 0 (does not interfere) to 10 (completely interferes).
Time Frame: Baseline, Week 3, Week 6, 1 month follow up, and 3 months follow up
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
Scores on a scale
  Pain interference at baseline | 1.73 [0.33 to 3.89]
  Pain interference at treatment week 3 | 3.00 [0.44 to 8.00]
  Pain interference at treatment week 6 | 6.70 [2.89 to 9.44]
  Pain interference at 1 month follow up | 3.17 [0 to 8.33]
  Pain interference at 3 months follow up | 1.87 [0 to 4.56]

15. Secondary Outcome: Mean Percentage Pain Relief After Medication
Description: The Brief Pain Inventory Scale questionnaire were used to assess pain relief after medication. Participants rated pain relief on a scale of 0% (no relief) to 100% (complete relief) and a mean and full range were reported.
Time Frame: Baseline, Week 3, Week 6, 1 month follow up, and 3 months follow up
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Full Range); unit: percentage pain relief
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
percentage pain relief
  Baseline | 90.0 [60 to 100]
  Treatment week 3 | 93.8 [85 to 100]
  Treatment week 6 | 44.0 [10 to 90]
  1 month follow up | 89.0 [75 to 100]
  3 months follow up | 83.0 [50 to 100]

16. Secondary Outcome: Duration of Overall Response (DOR)
Description: Duration of overall response is measured from the time measurement criteria are met for Complete Response until the first date that recurrent or progressive disease is objectively document. Complete Response was measured by the Response Evaluation Criteria in Solid Tumors (RECIST0 version 1.1. Complete Response is disappearance of all target lesions.
Time Frame: 12 months of follow up, approximately 14 months
Population: This outcome measure was not measurable.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
months | NA [NA to NA] — 1/6 participants enrolled withdrew before treatment. 1 participant never reached complete response. DOR was censored for all responders due to completion of follow up & median censoring time is 329 days. Median cannot be calculated as the median was not reached. A median cannot be reported unless 50% of participants have reached the endpoint. 50% did not reach the endpoint and came off study for complete follow-up.

17. Secondary Outcome: Percentage of Total Viable Cells That Were Cluster of Differentiation 3+ (CD3+) Cells in Biopsied Tissue
Description: Percentage of total viable cells that were Cluster of differentiation 3+ (CD3+) cells in biopsied tissue.
Time Frame: Baseline and 1 year
Population: 1/6 participants enrolled withdrew before treatment. 3 participants underwent optional biopsy.
Measure: Mean (Full Range); unit: percentage of cells
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 3
percentage of cells
  Baseline | 7.93 [5.69 to 9.1]
  1 year | 4.40 [2.4 to 5.7]

18. Secondary Outcome: Absolute Number of Cluster of Differentiation 3+ (CD3) Cells Per Gram of Biopsied Intestinal Tissue
Description: Absolute number of Cluster of differentiation 3+ (CD3) cells per gram of biopsied intestinal tissue. The number of CD3 positive cells were analyzed with flow cytometry of cellular suspensions from biopsy tissue.
Time Frame: Baseline and 1 year follow up
Population: 1/6 participants enrolled withdrew before treatment. 3 participants underwent optional biopsy.
Measure: Mean (Full Range); unit: CD3+cells/gm tissue(x 10^5)
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 3
CD3+cells/gm tissue(x 10^5)
  Baseline | 22.98 [12.1 to 29.3]
  1 year follow up | 13.62 [5.94 to 21.6]

19. Secondary Outcome: Number of Cluster of Differentiation 8+ (CD8) Cells Per Gram of Biopsied Intestinal Tissue
Description: Number of Cluster of differentiation 8+ (CD8) cells per gram of biopsied intestinal tissue. The number of CD8 positive cells were analyzed with flow cytometry of cellular suspensions from biopsy tissue.
Time Frame: Baseline and 1 year follow up
Population: 1/6 participants enrolled withdrew before treatment. 3 participants underwent optional biopsy.
Measure: Mean (Full Range); unit: CD8+cells/gm tissue(x 10^5)
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 3
CD8+cells/gm tissue(x 10^5)
  Baseline | 4.8 [1.4 to 5.6]
  1 year follow up | 4.0 [1.77 to 5.58]

20. Secondary Outcome: Number of Cluster of Differentiation 4+ (CD4) Cells Per Gram of Biopsied Intestinal Tissue
Description: Number of Cluster of Differentiation 4+ (CD4) cells per gram of biopsied intestinal tissue. The number of CD4 positive cells were analyzed with flow cytometry of cellular suspensions from biopsy tissue.
Time Frame: Baseline and 1 year follow up
Population: 1/6 participants enrolled withdrew before treatment.
Measure: Mean (Full Range); unit: CD4+cells/gm tissue(x 10^5)
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 5
CD4+cells/gm tissue(x 10^5)
  Baseline | 17.64 [9.54 to 23.2]
  1 year follow up | 12.72 [3.5 to 14.5]

21. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus (HIV) in Biopsy Tissue From Rectal Mucosa
Description: Optional snag biopsies pre and post were collected from participants rectal mucosa to enumerate cell counts.
Time Frame: Baseline and Course 1 Day 28
Population: This outcome measure could not be completed. 1/6 participants enrolled withdrew before treatment. No participants with HIV ribonucleic acid (RNA) underwent optional biopsy. HIV RNA is not analyzed unless a patient has HIV. Thus, data not collected.
Arm/Group | 1/Chemo + Radiation
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately, 36 months and 10 days.
Description: 1/6 participants enrolled withdrew before treatment.
Arm/Group | 1/Chemo + Radiation
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Chemo + Radiation (N=5)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Febrile neutropenia (Investigations) | 2 (2)
Fever (General disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1/Chemo + Radiation (N=5)
Abdominal pain (Gastrointestinal disorders) | 2 (4)
Alanine aminotransferase increased (Investigations) | 4 (7)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1)
Anal pain (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 4 (8)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Chills (General disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 5 (19)
Diarrhea (Gastrointestinal disorders) | 4 (14)
Dizziness (Nervous system disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ejaculation disorder (Reproductive system and breast disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Fatigue (General disorders) | 5 (8)
Fecal incontinence (Gastrointestinal disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (5)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, Tongue deviation (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (8)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Lymphocyte count decreased (Investigations) | 5 (34)
Memory impairment (Nervous system disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (8)
Neutrophil count decreased (Investigations) | 5 (15)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (2)
Perineal pain (Reproductive system and breast disorders) | 2 (4)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Clamminess (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) — - Other, Rash follicular, in and out of radiation and MTS-01 area
Skin and subcutaneous tissue disorders - Other, carbunkle (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Syncope (Nervous system disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Urinary tract pain (Renal and urinary disorders) | 4 (7)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
White blood cell decreased (Investigations) | 5 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-06): https://cdn.clinicaltrials.gov/large-docs/41/NCT01324141/Prot_SAP_000.pdf
  • Informed Consent Form (2014-04-02): https://cdn.clinicaltrials.gov/large-docs/41/NCT01324141/ICF_001.pdf